CLINICAL TRIAL: NCT04150341
Title: A Randomized, Double-blind, Placebo-controlled, 3-period Crossover Study to Evaluate the Effects of Repeated Doses of Inhaled TD-8236 and Impact on Airway Responses Following Allergen Challenge in Patients With Asthma
Brief Title: Effect of Inhaled TD-8236 on Allergen-induced Asthmatic Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0178; 2019-002915-24 (EudraCT Number)
Record Dates: First submitted 2019-10-15; First posted 2019-11-04 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-02

CONDITIONS: Asthma
Keywords: TD-8236; Asthma; Proof of concept
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- TD-8236 Dose A (low dose) (Experimental): TD-8236 Dose A (QD x 14 days)
  Interventions: Drug: TD-8236
- TD-8236 Dose B (high dose) (Experimental): TD-8236 Dose B (QD x 14 days)
  Interventions: Drug: TD-8236
- Placebo (Placebo Comparator): Placebo (QD x 14 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TD-8236 — The study drug will be administered by inhalation in the morning for 14 days during each period. A washout period of at least 21 days will exist between subsequent periods.
  Arms: TD-8236 Dose A (low dose); TD-8236 Dose B (high dose)
Drug: Placebo — The placebo will be administered by inhalation in the morning for 14 days during each period. A washout period of at least 21 days will exist between subsequent periods.
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, placebo-controlled study. The study will use a three-period, six-sequence, complete-block, cross-over study design to characterize two doses of inhaled TD-8236 compared to placebo in subjects with mild asthma and a known response to an allergen. Each of the three periods will be 14 days, followed by a washout period before the next period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age
* Willing and able to give informed consent and comply with study requirements
* Documented physician-diagnosed asthma for ≥ 4 months prior to Screening
* Body mass index (BMI) ≥ 18.0 and ≤ 35.0 kg/m2 at Screening and weighs ≥ 50 kg at Screening.
* Women of child bearing potential must have a negative pregnancy test
* Males and females must use a highly efficient birth control method
* Pre-bronchodilator FEV1 ≥ 70% predicted
* Documented allergy to at least one common allergen
* Dual responder to inhaled bronchial challenges
* Additional inclusion criteria apply

Exclusion Criteria:

* Positive for hepatitis A, B or C, HIV or tuberculosis
* Clinically significant abnormalities of laboratory evaluations
* Have abnormal ECG measurements
* Any sign of respiratory tract infection within 6 weeks of screening
* Have a current bacterial, parasitic, fungal or viral infection
* History of life-threatening asthma
* Uses or have used tobacco or nicotine-containing products within 6 months prior to screening
* Additional exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-08-28 (Actual); Study Completion 2020-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (2):
- United Kingdom (2):
  - Theravance Biopharma Investigational Site, London
  - Theravance Biopharma Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 participants were enrolled at 2 sites in the United Kingdom.
Pre-assignment Details: Participants were screened with an allergen challenge test within 35 days prior to first dosing. Participants received increasing concentrations of inhaled allergen until a decrease of ≥20% from preallergen forced expiratory volume (in 1 second) (FEV1) was observed during the 30 minutes following the most recent inhalation, and then monitored for a late asthmatic response (LAR).
Groups:
- TD-8236 150 mcg/TD-8236 1500 mcg/Placebo: Participants received TD-8236 150 mcg first, then TD-8236 1500 mcg, and then Placebo.
  All treatment periods were 14 days with a 21 day washout period between treatments.
- TD-8236 150 mcg/Placebo/TD-8236 1500 mcg: Participants received TD-8236 150 mcg first, then Placebo, and then TD-8236 1500 mcg.
  All treatment periods were 14 days with a 21 day washout period between treatments.
- Placebo/TD-8236 1500 mcg/TD-8236 150 mcg: Participants received Placebo first, then TD-8236 1500 mcg, and then TD-8236 150 mcg.
  All treatment periods were 14 days with a 21 day washout period between treatments.
- Placebo/TD-8236 150 mcg/TD-8236 1500 mcg: Participants received Placebo first, then TD-8236 150 mcg, and then TD-8236 1500 mcg.
  All treatment periods were 14 days with a 21 day washout period between treatments.
- TD-8236 1500 mcg/Placebo/TD-8236 150 mcg: Participants received TD-8236 1500 mcg first, then Placebo, and then TD-8236 150 mcg.
  All treatment periods were 14 days with a 21 day washout period between treatments.
- TD-8236 1500 mcg/TD-8236 150 mcg/Placebo: Participants received TD-8236 1500 mcg first, then TD-8236 150 mcg, and then Placebo.
  All treatment periods were 14 days with a 21 day washout period between treatments.
Period: Overall Study
Arm/Group | TD-8236 150 mcg/TD-8236 1500 mcg/Placebo | TD-8236 150 mcg/Placebo/TD-8236 1500 mcg | Placebo/TD-8236 1500 mcg/TD-8236 150 mcg | Placebo/TD-8236 150 mcg/TD-8236 1500 mcg | TD-8236 1500 mcg/Placebo/TD-8236 150 mcg | TD-8236 1500 mcg/TD-8236 150 mcg/Placebo
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 3 | 4
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized to 1 of 6 treatment sequences. Each treatment period was 14 days with a 21 day washout between treatments. All participants were randomized to receive all study drugs.
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Change From Baseline in Forced Expiratory Volume (in 1 Second) (FEV1) From 3 to 8 Hours After Inhaled Allergen Challenge at Day 14
Description: Values are reported as a weighted mean derived by calculating the AUC change from baseline over the relative time interval, divided by the time interval.
Time Frame: Day 14 of treatment period: 3 to 8 hours after allergen challenge
Population: Only participants with quantifiable measurements are included here.
Measure: Least Squares Mean (Standard Error); unit: liters
Groups:
- Placebo: Participants were administered inhaled doses of placebo matching TD-8236 once per day (QD) by dry powder inhaler on Day 1 to Day 14 of the 14 day treatment period. An allergen challenge was performed 1 hour after dosing on Day 14 at the dose of allergen required to achieve a successful response at screening.
- TD-8236 150 mcg: Participants were administered 150 microgram (mcg) inhaled doses of TD-8236 once per day (QD) by dry powder inhaler on Day 1 to Day 14 of the 14 day treatment period. An allergen challenge was performed 1 hour after dosing on Day 14 at the dose of allergen required to achieve a successful response at screening.
- TD-8236 1500 mcg: Participants were administered 1500 microgram (mcg) inhaled doses of TD-8236 once per day (QD) by dry powder inhaler on Day 1 to Day 14 of the 14 day treatment period. An allergen challenge was performed 1 hour after dosing on Day 14 at the dose of allergen required to achieve a successful response at screening.
Arm/Group | Placebo | TD-8236 150 mcg | TD-8236 1500 mcg
Number analyzed (Participants) | 22 | 22 | 20
liters | -0.53 (0.077) | -0.54 (0.077) | -0.57 (0.079)
Statistical Analysis 1: Comparison: Placebo vs TD-8236 150 mcg; Test type: Superiority; p = 0.881, Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.14 to 0.12]
Statistical Analysis 2: Comparison: Placebo vs TD-8236 1500 mcg; Test type: Superiority; p = 0.575, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.17 to 0.1]

2. Secondary Outcome: Area Under the Curve of Percentage Change From Baseline in Forced Expiratory Volume (in 1 Second) (FEV1) From 3 to 8 Hours After Inhaled Allergen Challenge at Day 14
Description: Values are reported as a weighted mean derived by calculating the AUC percentage change from baseline over the relative time interval, divided by the time interval.
Time Frame: Day 14 of treatment period: 3 to 8 hours after allergen challenge
Population: Only participants with quantifiable measurements are included here.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | TD-8236 150 mcg | TD-8236 1500 mcg
Number analyzed (Participants) | 20 | 22 | 22
percentage change | -16.92 (2.512) | -17.50 (2.516) | -17.97 (2.562)

3. Secondary Outcome: Maximum Decline in Forced Expiratory Volume (in 1 Second) (FEV1) From 3 to 8 Hours After Inhaled Allergen Challenge at Day 14
Time Frame: Day 14 of treatment period: 3 to 8 hours after allergen challenge
Population: Only participants with available data are included.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | TD-8236 150 mcg | TD-8236 1500 mcg
Number analyzed (Participants) | 22 | 22 | 20
liters | -0.83 (0.082) | -0.86 (0.082) | -0.85 (0.084)

4. Secondary Outcome: Maximum Percentage Decline in Forced Expiratory Volume (in 1 Second) (FEV1) From 3 to 8 Hours After Inhaled Allergen Challenge at Day 14
Time Frame: Day 14 of treatment period: 3 to 8 hours after allergen challenge
Population: Only participants with available data are included.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | TD-8236 150 mcg | TD-8236 1500 mcg
Number analyzed (Participants) | 22 | 22 | 20
percentage change | -27.02 (2.790) | -28.18 (2.794) | -26.88 (2.843)

5. Secondary Outcome: Area Under the Concentration-time Curve Over One 24-hour Dosing Interval (AUC0-24) of TD-8236 in Plasma
Time Frame: Day 14 of treatment period: Pre-dose and 0.5, 1, 2, 4, 6, 8 and 24 hours post-dose
Population: Only participants with quantifiable measurements are included here.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | TD-8236 150 mcg | TD-8236 1500 mcg
Number analyzed (Participants) | 4 | 20
h*ng/mL | 0.482 (48.8) | 1.54 (70.6)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of TD-8236 in Plasma During Dosing Interval
Time Frame: Day 14 of treatment period: Pre-dose and 0.5, 1, 2, 4, 6, 8 and 24 hours post-dose
Population: Only participants with quantifiable measurements are included here.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TD-8236 150 mcg | TD-8236 1500 mcg
Number analyzed (Participants) | 21 | 21
ng/mL | 0.0207 (46.4) | 0.160 (54.3)

7. Secondary Outcome: Time to Maximum Observed Concentration (Tmax) of TD-8236 in Plasma Over a Dosing Interval
Time Frame: Day 14 of treatment period: Pre-dose and 0.5, 1, 2, 4, 6, 8 and 24 hours post-dose
Population: Only participants with quantifiable measurements are included here.
Measure: Median (Full Range); unit: hours
Arm/Group | TD-8236 150 mcg | TD-8236 1500 mcg
Number analyzed (Participants) | 21 | 21
hours | 0.950 [0.483 to 1.03] | 0.550 [0.467 to 1.07]

8. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any adverse event (AE) that begins on or after the date of first dose of study drug up to the date of last dose of study drug plus the number of days in the follow-up period.
  The severity of TEAEs were also assessed and were classified as mild, moderate or severe per the definitions below:
  Mild - The AE is noticeable to the participant and/or the investigator, but does not interfere with routine activity.
  Moderate - The AE interferes with routine activity, but responds to symptomatic therapy or rest.
  Severe - The AE significantly limits the participant's ability to perform routine activities despite symptomatic therapy.
Time Frame: Day 1 to end of follow-up (up to approximately 98 days)
Population: Only participants with available data are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TD-8236 150 mcg | TD-8236 1500 mcg
Number analyzed (Participants) | 24 | 23 | 24
Participants
  Any TEAE | 10 | 9 | 9
  Moderate or Severe TEAE | 3 | 3 | 2

ADVERSE EVENTS:
Time Frame: Day 1 to end of follow-up (up to approximately 98 days)
Arm/Group | Placebo | TD-8236 150 mcg | TD-8236 1500 mcg
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 10/24 | 9/23 | 9/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | TD-8236 150 mcg (N=23) | TD-8236 1500 mcg (N=24)
Exposure to SARS-CoV-2 (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Forced expiratory volume decreased (Investigations) | 1 (1) | 1 (2) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 5 (7) | 4 (5)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT04150341/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04150341/SAP_001.pdf